CLINICAL TRIAL: NCT06145204
Title: Effect of Complex Decongestive Therapy and Correlation Between Volume and Pain in Lower Limb Lymphedema: a Prospective Study
Brief Title: Correlation Between Volume and Pain in Lower Limbs Lymphoedema
Status: Completed | Type: Observational
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Deltombe Thierry, Professeur clinique, University Hospital of Mont-Godinne
Other Study IDs: B0392022000072
Record Dates: First submitted 2023-08-07; First posted 2023-11-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Lymphedema, Lower Limb
Keywords: pain; volume; adult
MeSH Terms: conditions — Lymphedema; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- single-group: Adult patients suffering from lymphoedema of one or both lower limbs, capable of expressing their wishes and cared for their pathology at the Godinne Lymphoedema Reference Center.
  There is no intervention (observational study). Questionnaires will be given at the beginning (Day 0) and the end (Day 4) of the cure and at the start of next cure (Month 3 to 8) : Lymph-iCf-LL, OMSPQ, BPI-sf.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — anamnesis, OMSPQ, Brief Pain Inventory-short form, lymph-ICF-LL

SUMMARY:
The vascular physiotherapy department of the UCL University Clinics of Mont-Godinne specializes in the physiotherapeutic management of lymphoedema. Since 2018, an agreement has been established with INAMI to evaluate the effect of complex decongestion therapy on lymphoedema and its impact on patients' quality of life.

One of the aims of the treatment is to reduce the volume of lymphoedema and the discomfort or even pain associated with it. More generally, pain can have a significant functional impact, especially when it becomes chronic. As pain is subjective and influenced by many factors, it is difficult to assess it. Therefore it is interesting to consider psychosocial factors when assessing pain, in order to propose a global management approach.

At Mont-Godinne, pain-related data is currently collected on a numerical scale from 0 to 10, using the Lymph-ICF questionnaire. Moreover, in Belgium, reimbursement for lymphoedema care in the form of pathology E or F is based mainly on volume measurements.

The main aim of this study is to identify correlations between lymphoedema volume and pain related to lower limbs and to determine if pain could reduced when lymphoedema volume is decreased using current therapy. The second objective is collecting demographic data to assess the need for a comprehensive, specific and systematic approach to pain in the management of lymphoedema.

To proceed this assessment, we have sought the opinion of the Ethics Committee regarding the anonymous collection of new data from patients treated via a medical history and the introduction of two validated questionnaires (Brief Pain Inventory - short version and Orebro Musculoskeletal Pain Screening Questionnaire (OMSPQ) - short version) at D0 (start of complex decongestion therapy), D4 (end of complex decongestion therapy) and M3-8 (start of next complex decongestion therapy). No interventions or measures other than those used in clinical practice will be added.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients with lymphoedema of one or both lower limbs diagnosed by three-stage lymphoscintigraphy, or clinically if it is medically impossible to perform three-stage lymphoscintigraphy for good reason.

Exclusion Criteria:

* Patient under 18 years of age
* Pain not related to lymphoedema
* Inability to read and understand French to answer questionnaires
* Patient with infection of the lower limb(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from lymphoedema of one or both lower limbs, capable of expressing their wishes and cared for at the Godinne Lymphoedema Reference Center.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
pain assessment using questionnaires: Lymph-iCf-LL | at the beginning (Day 0) and the end (Day 4) of the cure
  we will compare the results in % between the beginning and the end of the cure
pain assessment using questionnaires: OMSPQ | at the beginning (Day 0) and the end (Day 4) of the cure and at the beginning of the next cure (Month 3 to 8)
  we will compare the results in % between the beginning and the end of the cure and the beginning of the next cure
pain assessment using questionnaires: BPI-sf | at the beginning (Day 0) and the end (Day 4) of the cure and at the beginning of the next cure (Month 3 to 8)
  we will compare the results between the beginning and the end of the cure and the beginning of the next cure with two scores: intensity and interference score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU UCL Namur site Godinne, Yvoir, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No